CLINICAL TRIAL: NCT00006056
Title: Pilot Study of Unrelated Donor Hematopoietic Stem Cell Transplantation in Patients With Life Threatening Hemophagocytic Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fairview University Medical Center (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/15106; UMN-MT-1997-08; UMN-MT-9708
Record Dates: First submitted 2000-07-05; First posted 2000-07-06 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-10

CONDITIONS: Chediak-Higashi Syndrome; Graft Versus Host Disease; X-Linked Lymphoproliferative Syndrome; Familial Erythrophagocytic Lymphohistiocytosis; Hemophagocytic Lymphohistiocytosis; Virus-Associated Hemophagocytic Syndrome
Keywords: Chediak-Higashi syndrome; X-linked lymphoproliferative syndrome; disease-related problem/condition; familial erythrophagocytic lymphohistiocytosis; genetic diseases and dysmorphic syndromes; graft versus host disease; hematologic disorders; hemophagocytic lymphohistiocytosis; histiocytosis; immunologic disorders and infectious disorders; primary immunodeficiency disease; rare disease; virus-associated hemophagocytic syndrome
MeSH Terms: conditions — Chediak-Higashi Syndrome; Graft vs Host Disease; Lymphoproliferative Disorders; Lymphohistiocytosis, Hemophagocytic; Genetic Diseases, Inborn; Hematologic Diseases; Histiocytosis; Immune System Diseases; Communicable Diseases; Primary Immunodeficiency Diseases; Rare Diseases | interventions — Antilymphocyte Serum; Busulfan; Cyclophosphamide; Cyclosporine; Etoposide; Filgrastim; Methotrexate

INTERVENTIONS:
Drug: anti-thymocyte globulin
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: etoposide
Drug: filgrastim
Drug: methotrexate
Procedure: allogeneic hematopoietic stem cell transplantation

SUMMARY:
OBJECTIVES: I. Determine the efficacy of unrelated donor hematopoietic stem cell transplantation in the treatment of patients with life threatening hemophagocytic disorders.

II. Determine the rate of disease free survival, incidence of graft failure, and incidence of graft versus host disease in these patients after undergoing this treatment regimen.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive oral busulfan twice a day on days -9 to -6; cyclophosphamide IV over 1 hour on days -5 to -2; etoposide IV over 4 hours on days -5 to -3; and anti-thymocyte globulin IV twice a day on days -2 and -1 and days 1 and 2. Patients undergo allogeneic hematopoietic stem cell transplantation on day 0. Filgrastim (G-CSF) is administered subcutaneously beginning on day 1 and continuing until blood counts recover. Patients receive graft versus host disease prophylaxis with methotrexate IV on days 1, 3, 6, and 11 and cyclosporine IV over 1-4 hours (orally once the patients resumes eating) every 12 hours (every 8 hours for pediatric patients) starting on or prior to day -3 and continuing up to 1 year.

Patients are followed at days 28 and 100, at 6 months and 1 year, and then annually for 5 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Patients diagnosed with any of the following active but stable, or nonactive/quiescent, hemophagocytic disorders:

* Hemophagocytic lymphohistiocytosis (HLH)
* Fever greater than 38.5 degrees Celsius
* Splenomegaly (greater than 3 cm below costal margin)
* Hemophagocytosis in bone marrow or spleen or lymph nodes
* Disease may be confirmed by positive family history
* No evidence of malignancy
* Hypertriglyceridemia and/or hypofibrinogenemia
* Fasting triglycerides at least 2.0 mmol/L or at least 3 standard deviations above normal for age
* Fibrinogen no greater than 1.5 g/L or no greater than 3 standard deviations above normal
* Cytopenia (affecting at least 2 of 3 lineages in the peripheral blood)
* Hemoglobin less than 9.0 g/L
* Platelet count less than 100,000/mm3

X-linked lymphoproliferative disorder (XLP)

Two or more maternally related males manifesting at least one of the following XLP phenotypes:

* Fulminant infectious mononucleosis
* Dysgammaglobulinemia
* Malignant lymphoma/lymphoproliferative disorder
* Aplastic anemia
* Lymphoid granulomatosis/vasculitis OR
* A maternally related male in an established XLP kindred who has strong genetic (RFLP) linkage to the XLP locus

Chediak-Higashi syndrome

Partial oculocutaneous albinism (hair, skin, eyes)

Frequent bacterial infections

Large peroxidase positive granules in leukocytes of peripheral blood or bone marrow

Positive family history or parental consanguinity is supportive of the diagnosis

May not have entered accelerated phase as defined by any of the following:

* Lymphadenopathy
* Pancytopenia
* Histiocytes with hemophagocytosis in bone marrow, lymph nodes, liver, or spleen

Viral associated hemophagocytic syndrome (VAHS)

Relapsed after prior therapy or supportive care

Diagnostic criteria as for HLH

No hemophagocytic disorders secondary to underlying malignancy

Patients 35 years of age and under must have a hematopoietic stem cell donor that is one of the following:

* HLA A and B identical OR
* Single HLA A or B serologic mismatch with DRB1 identity OR
* HLA A or B serologic identity with a single DRB1 mismatch

Patients 36 to 55 years of age must have a hematopoietic stem cell donor that is one of the following:

* HLA A and B and HLA DRB1 identical OR
* Single HLA A or B serologic mismatch with DRB1 identity

Patients receiving umbilical cord blood must have an unrelated donor with no more than two antigen HLA A, B, or DRB1 mismatches

--Patient Characteristics--

Performance status: Karnofsky 70-100% OR Age less than 16 years: Lansky 50-100%

Life expectancy: Not severly limited by another disease

Hepatic: SGOT less than 3 times normal Bilirubin less than 2.5 mg/dL

Renal: Creatinine normal OR Creatinine clearance or glomerular filtration rate greater than 50% normal

Cardiovascular: If symptomatic, ventricular ejection fraction must be greater than 40% and must improve with exercise OR Shortening fraction normal on echocardiogram

Pulmonary:

* If symptomatic, DLCO greater than 45% predicted (corrected for hemoglobin)
* In children unable to perform pulmonary function testing, oxygen saturation must be greater than 95%

Other: HIV negative No significant active infections

Ages: 0 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2000-03

CONTACTS AND LOCATIONS:
Overall Officials: K. Scott Baker, Study Chair — Fairview University Medical Center
Locations (1):
- Fairview University Medical Center, Minneapolis, Minnesota, United States